CLINICAL TRIAL: NCT01625221
Title: An Observational Clinical Feasibility Study of The Magnetic Anal Sphincter
Brief Title: Feasibility Study of the Magnetic Anal Sphincter (FENIX System)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1876, 1990, 2321
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Fecal Incontinence
Keywords: FENIX
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic anal sphincter augmentation (Experimental): The implantable single-use Magnetic Anal Sphincter (FENIX) device consists of a series of titanium beads with magnetic cores that are linked together with independent titanium wires forming an annular shape. The device is supplied sterile and is placed through an open incision.
  Interventions: Device: Magnetic Anal Sphincter

INTERVENTIONS:
Device: Magnetic Anal Sphincter — The implantable single-use Magnetic Anal Sphincter (FENIX) device consists of a series of titanium beads with magnetic cores that are linked together with independent titanium wires forming an annular shape. The device is supplied sterile and is placed through an open incision.

SUMMARY:
The purpose of this feasibility study is to obtain preliminary safety and effectiveness information and develop procedural optimization for the Magnetic Anal Sphincter device (FENIX System) in reinforcement of anal sphincter function to treat severe fecal incontinence (FI).

DETAILED DESCRIPTION:
Study subjects followed to 12 months post implant outside the U.S. Study subjects followed to 5 years post implant in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years, <85 years, life expectancy >3yrs.
* Documented history of severe fecal incontinence for at least 6 months
* Subject diary documents ≥ 2 episodes per week on average over diary period, leakage greater than seepage
* Subject has failed standard conservative and medical therapy
* Subject is a surgical candidate.
* Subject is willing and able to cooperate with follow-up examinations.
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form and provided authorization to use and disclose information for research purposes.

Exclusion Criteria:

* Subject has history of significant obstructed defecation or other significant chronic defecatory motility disorders
* Subject has current, external full thickness rectal prolapse or vaginal prolapse
* Subject has an electric or metallic implant within 10cm of the area of device placement
* Subject has Inflammatory Bowel Disease
* Subject has Irritable Bowel Syndrome
* Subject has systemic disease as source of FI (scleroderma, neurologic disorders, Crohn's)
* Subject has active pelvic infection
* Subject has chronic diarrhea
* Subject diagnosed with anal, rectal, or colon cancer within 2 years
* Subject has had prior anterior resection of the rectum
* Subject has undergone pelvic radiation therapy
* Subject has significant scarring of the recto-vaginal septum, a permanent implant in the recto-vaginal septum, or a history of recto-vaginal fistula
* Subject has had previous anorectal posterior compartment surgery
* The procedure is an emergency procedure
* Subject is currently being treated with another investigational drug or investigational device.
* Subject cannot understand trial requirements or is unable to comply with follow-up schedule.
* Subject is pregnant or nursing, or plans to become pregnant.
* Subject has history of complex anal fistula

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Colon and Rectal Surgery Associates, Minneapolis, Minnesota
  - Providence Medical Research Center, Spokane, Washington
- Arhus Universitetshospital, Aarhus, Denmark
- University of Medicine, Nantes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnetic Anal Sphincter Augmentation
Started | 35
Completed | 28
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Anal Sphincter Augmentation
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 1
Region of Enrollment [Number; unit: participants]
  France | 15
  United States | 15
  Denmark | 5
Fecal incontinence episodes [Mean (Standard Deviation); unit: episodes per week] | 13.9 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The safety objective will be met via reporting all adverse events at various time points including implant, 6 weeks, 3 months, 6 months, and 12 months (and then semi-annually until 5 years post-implant at U.S. sites). Serious device- and procedure-related adverse events will be summarized separately. Safety will be characterized by physical examination and pelvic X-ray evaluations.
Time Frame: 60 months
Population: All adverse events as reported by investigators
Measure: Number; unit: Number of events
Arm/Group | Magnetic Anal Sphincter Augmentation
Number analyzed (Participants) | 35
Number of events
  All Adverse Events | 223
  Serious Device or Procedure-related Adverse Events | 7

2. Primary Outcome: Reduction in Fecal Incontinence Symptoms
Description: Effectiveness will be characterized as the reduction of FI symptoms by subjective measurements using the FISI, Wexner, and FIQOL scores and a three week diary documenting episodes of incontinence.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Magnetic Anal Sphincter Augmentation
Number analyzed (Participants) | 28
episodes per week | 3.8 (5.1)

ADVERSE EVENTS:
Arm/Group | Magnetic Anal Sphincter Augmentation
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 12/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magnetic Anal Sphincter Augmentation (N=35)
Infection (Infections and infestations) | 4
Device erosion (Skin and subcutaneous tissue disorders) | 1
Impaction or defecatory disorder (Gastrointestinal disorders) | 1
Allergy, inflammation reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magnetic Anal Sphincter Augmentation (N=35)
Device erosion (Skin and subcutaneous tissue disorders) | 3
Pain (Gastrointestinal disorders) | 6
Impaction or defecatory disorder (Gastrointestinal disorders) | 2
Rectal bleeding (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days